CLINICAL TRIAL: NCT03369158
Title: A Prospective Clinical Survey on Accuracy of Pedicle Screws Positioning With MySpine Versus Free Hand Technique
Brief Title: Pedicle Screw Positioning With MySpine vs Free Hand Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05.005.01
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2017-11

CONDITIONS: Spinal Deformity

ARMS (2):
- MySpine (Experimental): Patients operated for spinal stabilization through patient specific pedicle screw guide "MySpine"
  Interventions: Procedure: patient specific pedicle screw positioning guide; Device: MUST pedicle screw
- Free hand technique (Active Comparator): Patients operated for spinal stabilization through standard free hand technique
  Interventions: Procedure: Free hand technique pedicle screw positioning; Device: MUST pedicle screw

INTERVENTIONS:
Procedure: patient specific pedicle screw positioning guide
  Other Names: MySpine
  Arms: MySpine
Procedure: Free hand technique pedicle screw positioning
  Arms: Free hand technique
Device: MUST pedicle screw

SUMMARY:
Randomized clinical study in order to evaluate the accuracy of pedicle screw positioning during spine surgery performed with MySpine patient match positioning guide or Free hand technique.

DETAILED DESCRIPTION:
The proposed study seeks to assess the intraoperative accuracy of the Medacta patient-specific MySpine® pedicle screws placement guides in comparison to free-hand technique.

A pre-operative CT scan of the spine is obtained to create a 3-dimensional model of the patient's spine for the MySpine patient group. This model is then used to preoperatively plan the patient's surgery implantation itself, with the same goals of both free-hand and computer assisted techniques. The theoretical advantage of this technique is accurate implant placement without the added surgical time and complexity of the procedure, with lower radiation exposure thanks to less steps of fluoroscopy checks.

The hypothesis for the present study is that the MySpine® technique can place pedicle screws more accurately in comparison to free-hand technique.

The accuracy of the final implant position with respect to the pre-operative planning will be evaluated through CT post-op analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 12 years
* patients suffering from coronal or sagittal spinal deformities that will undergo a surgical treatment with a posterior approach and pedicle screws placement
* Patients suitable to undergo spinal stabilization (according to the label indication/contraindications)
* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained when indication to surgery is confirmed.

Exclusion Criteria:

* Patient with congenital spinal deformity (emeverebre, vertebra wedge, vertebrate butterfly, congenital bar, vertebra block)
* Patients with a previous fusion of the spine in the region where screws will be inserted
* Patients with any allergy to the device implanted
* Patients who will be not able to provide their written consent to the study participation
* Patients who are incapable of understanding and wanting

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2017-02-13 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- MySpine: Patients operated for spinal stabilization through patient specific pedicle screw guide "MySpine"
  patient specific pedicle screw positioning guide
  MUST pedicle screw
- Free Hand Technique: Patients operated for spinal stabilization through standard free hand technique
  Free hand technique pedicle screw positioning
  MUST pedicle screw
Period: Overall Study
Arm/Group | MySpine | Free Hand Technique
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MySpine | Free Hand Technique | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (15.3) | 26 (17.2) | 31 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Pedicle Screw Positioning
Description: Pedicle screw accuracy is defined as having the entire screw contained within the cortices of each respective pedicle.
Time Frame: 1 week after surgery
Measure: Number (95% Confidence Interval); unit: percentage of screw
Units Other Than Participants: screw
Arm/Group | MySpine | Free Hand Technique
Number analyzed (Participants) | 14 | 15
Number analyzed (screw) | 297 | 243
percentage of screw | 90.24 [86.86 to 93.6] | 83.13 [78.42 to 87.84]

2. Secondary Outcome: Radiological Evaluation of Pedicle Screw Malposition
Description: A CT will be performed before discharge to evaluate the severity of pedicle screws malposition according to Gertzbein in grades 0, A, B or C, with grades 0 or A considered as "safe area.". Level 0 (perfect corrected positioning of the screw), level A (0-2 mm of violation), level B (2-4 mm of violation), level C (˃4mm of violation). The better outcomes correspond to level 0 and the worst to level C.
Time Frame: 1 weeks after surgery
Measure: Count of Units; unit: screws
Units Other Than Participants: screws
Arm/Group | MySpine | Free Hand Technique
Number analyzed (Participants) | 14 | 15
Number analyzed (screws) | 297 | 243
screws
  Group 0 | 224 | 160
  Group A | 44 | 42
  Group B | 16 | 19
  Group C | 13 | 22

3. Secondary Outcome: Occurrence of Malposition Side
Description: Evaluation of malposition on the medial or lateral side
Time Frame: 1 weeks after surgery
Measure: Number; unit: screws
Units Other Than Participants: screw
Arm/Group | MySpine | Free Hand Technique
Number analyzed (Participants) | 14 | 15
Number analyzed (screw) | 297 | 243
screws
  Lateral misplacement | 19 | 31
  Medial misplacement | 46 | 54

4. Secondary Outcome: Incidence of Adverse Event
Description: Occurrence of intra-operative complications reporting
Time Frame: intraoperatively, up to 1 week after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MySpine | Free Hand Technique
Number analyzed (Participants) | 14 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | MySpine | Free Hand Technique
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No